CLINICAL TRIAL: NCT02810301
Title: A Randomized, Double-Blind, Placebo-Controlled Study on the Efficacy of Bifidobacterium Longum Probiotic ES1 for the Treatment of Non-Celiac Gluten Sensitivity
Brief Title: Efficacy of Probiotic ES1 for the Treatment of Non-Celiac Gluten Sensitivity
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Exzell Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EX-ES01
Record Dates: First submitted 2016-06-17; First posted 2016-06-22 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Non-Celiac Gluten Sensitivity
Keywords: gluten; non-celiac; gluten sensitivity
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Probiotic ES1) (Experimental): Capsules containing 1 billion CFU of B. longum ES1 per capsule. One capsule taken before and after consuming 2 slices of bread for 7 days.
  Interventions: Other: Probiotic ES1
- Placebo (Placebo Comparator): Capsules not containing the active ingredient B. longum ES1. One capsule taken before and after consuming 2 slices of bread for 7 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Probiotic ES1 — B. longum ES1 is formulated for oral use as Glutagest. Each capsule contains 1 billion CFU of B. longum. The capsules are off-white in color and cylindrical in shape with approximate dimensions of 19 mm x 6.63 mm and a weight of 500 mg. Non-medicinal ingredients consist of the common excipients filler rice maltodextrin, lubricant stearic acid, and encapsulating agent vegetable cellulose.
  Other Names: Glutagest
  Arms: Treatment (Probiotic ES1)
Other: Placebo — The placebo is composed of the same non-medicinal ingredients as the investigational product (IP) (i.e. rice maltodextrin, stearic acid, and vegetable cellulose) but it does not contain the active ingredient B. longum ES1. The placebo is designed to resemble the IP in terms of physical appearance.
  Arms: Placebo

SUMMARY:
Study to demonstrate the efficacy of Probiotic ES1 in alleviating symptoms of gluten sensitivity in non-celiac gluten sensitive subjects exposed to a small, fixed amount of gluten.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study. Sixty non-celiac gluten sensitive subjects will be randomized into one of two groups; Probiotic ES1 or placebo. For the duration of the study, subjects must adhere to a gluten-free diet, apart from a scheduled fixed gluten exposure of two slices of bread once daily. Subjects will be required to take 1 capsule before and after consuming the two slices of bread and score the severity of their symptoms in a diary provided for the duration of the study (7 days).

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65
* Male or non-pregnant, non-lactating females.
* Documented or self-diagnosed gluten sensitivity that is well-controlled.
* Negative celiac serology to eliminate Celiac Disease at screening.
* Written informed consent prior to any screening procedure.
* Ability and willingness to comply with study requirements.
* Adherence to a gluten-free diet during period of the study and 1 week prior to the first dose.
* BMI < 35 kg/m2.

Exclusion Criteria:

* History of diagnosis of Celiac Disease.
* Positive pregnancy test at screening.
* Positive HIV, Hepatitis, or Tuberculosis infection.
* History of substance abuse within last 5 years.
* Alcohol consumption of > 2 standard drink equivalents per day.
* Recent myocardial infarction within past 3 months, recent stroke within past 12 months, recent abdominal surgery within past 12 months, history of any malignancies and/or active treatment for a psychiatric disorder.
* Use of systemic biologics within 6 months of the study.
* Use of oral probiotics within 2 weeks of the study.
* Use of NSAIDS or aspirin within 7 days of the study.
* Use of immunosuppressants within 30 days of the study.
* Family history (first degree relative) of Celiac Disease.
* Received an investigational product within 1 month of study.
* History of digestive enzyme deficiencies.
* History of severe reactions to low doses of gluten/accidental exposure to gluten.
* History of wheat allergy (positive reactions to the skin-prick test or the IgE blood test).
* History of lactose, milk protein and/or FODMAP allergies.
* Subjects who have an immune-compromised condition.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-12 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Change in mean overall symptoms (as assessed by a 100-mm visual analog scale) in active versus placebo. | Baseline to 7 days.
  The efficacy of Probiotic ES1 using a 100-mm visual analog scale (VAS).

SECONDARY OUTCOMES:
Adverse event assessment | Baseline to 7 days.
  The incidence and severity of adverse events.
Change in individual symptoms (as assessed by a 100-mm VAS) in active versus placebo. | Baseline to 7 days.
  The efficacy of Probiotic ES1 using a 100-mm visual analog scale (VAS).

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Pardeep Nijhawan, MD, Principal Investigator — Digestive Health Clinic / Exzell Pharma Inc.
Locations (1):
- Digestive Health Clinic Research, Richmond Hill, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided